CLINICAL TRIAL: NCT02659904
Title: The Quantitative Changes in Palatal Donor Sites Thickness After Free Gingival Graft Harvesting
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: İlker KESKINER (Other)
Responsible Party: Sponsor-Investigator, İlker KESKINER, Principal Investigator, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/103
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Healthy; Gingival Recession
Keywords: Free gingival graft; Palatal donor site healing
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Less than 2 mm (Active Comparator): Palatal mucosa thickness was measured from baseline to 1, 3 and 6 months after graft harvesting Intervention: Less than 2 mm remaining palatal tissue thickness
  Interventions: Other: Less than 2 mm remaining palatal tissue thickness
- 2 mm or more (Active Comparator): Palatal mucosa thickness was measured from baseline to 1, 3 and 6 months after graft harvesting Intervention: 2 mm or more remaining palatal tissue thickness
  Interventions: Other: 2 mm or more remaining palatal tissue thickness

INTERVENTIONS:
Other: Less than 2 mm remaining palatal tissue thickness — The greater palatine and incisive nerves were blocked with 2% lidocaine, 1:100,000 epinephrine injection. After preparation of the recipient bed, free gingival graft was harvested using a handle with knife at palatal donor side with acrylic stent guidance.
  Arms: Less than 2 mm
Other: 2 mm or more remaining palatal tissue thickness — The greater palatine and incisive nerves were blocked with 2% lidocaine, 1:100,000 epinephrine injection. After preparation of the recipient bed, free gingival graft was harvested using a handle with knife at palatal donor side with acrylic stent guidance.
  Arms: 2 mm or more

SUMMARY:
Our primary objective in this clinical intervention study, therefore, was to explored the effect of residual tissue thickness on the palatal mucosa healing from baseline to 1, 3 and 6 months after free gingival graft harvesting in order to determine as soon as possible to re-harvest gingival graft from same site.

DETAILED DESCRIPTION:
Forty individuals (19 males and 21 females; age range: 18-35 years) were enrolled in the study. Based on the remaining tissue at donor site after free gingival graft harvesting, individuals were divided into two groups: 1.0-1.9 millimeter (mm) remaining tissue at donor site after harvesting (n = 20), 2-2.9 mm remaining tissue at donor site after harvesting. Tissue filling in defect area from three points (mesial, central and distal) was measured at various time-points (baseline, post-operative 1, 3, 6 months).

ELIGIBILITY:
Inclusion Criteria:

* All individuals received oral hygiene instructions and full-mouth scaling was performed. -They were instructed to perform a non-traumatic brushing technique (Roll) using an ultra-soft toothbrush
* Individuals were re-evaluated at 8 weeks after initial therapy, and only full mounth plaque score and full mounth bleeding score <15% were enrolled to the surgical procedure
* mucogingival defects which for soft tissue graft application were indicated
* For Less than 2 mm group, between 2.5 and 3.4 mm palatal thickness at each measurement points before graft harvesting
* For 2 mm or more group, between 3.5 and 4.4 mm palatal thickness at each measurement points before graft harvesting.

Exclusion Criteria:

* periapical or palatal pathologies,
* absence teeth from canine to first molar,
* excessive forces including mechanical forces from orthodontics and occlusion,
* systemic diseases that would contraindicate for periodontal surgery or interfere with tissue healing, chronic high-dose steroid therapy, radiation or immunosuppressive therapy, pregnancy, lactation, smoking, or allergy or sensitivity to any drug
* Study participants had no history of drug therapy known to interfere with healing and to cause gingival enlargement
* Individuals who had complication such as bleeding, necrosis and delay healing during or after surgery were excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in remaining palatal tissue thickness | From baseline remaining palatal tissue thickness to post-operative 1, 3, 6 months

REFERENCES:
- [Derived] Keskiner I, Aydogdu A, Balli U, Kaleli AE. Quantitative changes in palatal donor site thickness after free gingival graft harvesting: a pilot study. J Clin Periodontol. 2016 Nov;43(11):976-984. doi: 10.1111/jcpe.12592. Epub 2016 Sep 9. PMID 27330024